CLINICAL TRIAL: NCT01247077
Title: Neuropsychologic and Immunological Evaluation in Treatment of Thyroid Diseases. Is Selenium Efficient?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jan Calissendorff, MD, Senior consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: DLL-159361
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: QoL Before and After 9 Month of Medical Treatment of Graves´Thyrotoxicosis; Potential Effect of Selenium
Keywords: selenium; neuropsychological testing; autoantibodies
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Active Comparator): Placebo and thyroxin + methimazole
  Interventions: Other: placebo
- selenium (Placebo Comparator): selenium + methimazole + thyroxin
  Interventions: Other: selenium

INTERVENTIONS:
Other: selenium — 200 ug selenium once daily
  Arms: selenium
Other: placebo
  Arms: placebo

SUMMARY:
Graves thyrotoxicosis is a common autoimmune disease. Patients suffer at diagnosis from weight loss, increased heart rate and stress intolerance. Some patients have difficulties in regaining quality of life. Diagnosis is found through elevated thyroid hormones thyroxin, suppressed TSH (thyroid stimulating hormone) from the pituitary and elevated stimulatory antibodies, TRAb (thyrotropin receptor antibody) to the thyroid. Selenium is sparse in western Europe. This compound has important function in thyroid hormone metabolism and on the immune system. It is not known whether addition of selenium affects the well being of patients with Graves´thyrotoxicosis. The subject of this study is to investigate this

DETAILED DESCRIPTION:
In the County of Södermanland we include 44 patients with Graves´thyrotoxicosis. They are treated with methimazole and thyroxin, and randomised to selenium or placebo. Neuropsychological investigation is performed, before medical treatment is commenced and repeated after 9 month. Serum concentration of thyroid hormon levels, autoantibodies and selenium are followed.

ELIGIBILITY:
Inclusion Criteria:

* New diagnose of autoimmune thyrotoxicosis
* biochemically proven with increased thyroxin
* low TSH and elevated TRAb/or positive scintigraphy.
* Age 18 - 55. Willing to participate -

Exclusion Criteria:

* No previous head trauma,
* No difficulties with swedish language,
* No medication which could affective neuropsychological testing,
* No planned or ongoing pregnancies.
* Normal intellectual capacity.
* No severe ophthalmopathy, or other severe disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Effect on neuropsychological well-being | Inclusion going on until the end of 2011

SECONDARY OUTCOMES:
Potential effect on autoantibodies | Inclusion for the rest of 2011

CONTACTS AND LOCATIONS:
Overall Officials: Jan Calissendorff, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Jan Calissendorff, Medical clinic, Eskilstuna, Sweden, Eskilstuna, Södermanland County
  - Emil Mikulski, Eskilstuna